CLINICAL TRIAL: NCT03795298
Title: Comparison of Anticoagulation With Left Atrial Appendage Closure After AF Ablation
Acronym: OPTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S2239
Record Dates: First submitted 2019-01-02; First posted 2019-01-07 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation; Left atrial appendage; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- WATCHMAN FLX (Experimental): WATCHMAN FLX implant including modified post-implant drug regimen.
  Interventions: Device: WATCHMAN FLX Implant
- Market-approved OAC (Active Comparator): Used per IFU for atrial fibrillation stroke prevention for the duration of the trial.
  Interventions: Drug: Market-approved OAC

INTERVENTIONS:
Device: WATCHMAN FLX Implant — Left atrial appendage closure with the WATCHMAN FLX device
  Arms: WATCHMAN FLX
Drug: Market-approved OAC — Used per IFU for atrial fibrillation stroke prevention for the duration of the trial.
  Arms: Market-approved OAC

SUMMARY:
The primary objective of this study is to determine if left atrial appendage closure with the WATCHMAN FLX Device is a reasonable alternative to oral anticoagulation following percutaneous catheter ablation for high risk patients with non-valvular atrial fibrillation.

DETAILED DESCRIPTION:
This study is a prospective, randomized, multi-center, global investigation to determine if left atrial appendage closure with the WATCHMAN FLX Device is a reasonable alternative to oral anticoagulation in patients after AF ablation.

A subject who signs informed consent is considered enrolled in the study. Subjects will be randomized to OAC or WATCHMAN FLX in equal fashion. Randomization will be stratified by sequential vs. concomitant planned ablation +/- WATCHMAN implantation, to help ensure balance of treatment assignments within the sequential and concomitant groups.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is of legal age to participate in the study per the laws of their respective geography.
2. Underwent a prior catheter ablation procedure for non-valvular AF between 90 and 180 days prior to randomization (sequential) or is planning to have clinically indicated catheter ablation within 10 days of randomization (concomitant).
3. The subject has a calculated CHA2DS2-VASc score of 2 or greater for males or 3 or greater for females.
4. The subject is deemed to be suitable for the defined protocol pharmacologic regimen.
5. The subject is able to undergo TEE examinations.
6. The subject or legal representative is able to understand and is willing to provide written informed consent to participate in the trial.
7. The subject is able and willing to return for required follow-up visits and examinations.

Exclusion Criteria:

1. The subject is currently enrolled in another investigational study that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance must be brought to the attention of the sponsor to determine eligibility, regardless of type of co-enrollment being proposed.
2. The subject requires long-term anticoagulation therapy for reasons other than AF-related stroke risk reduction, for example due to an underlying hypercoagulable state (i.e., even if the device is implanted, the subjects would not be eligible to discontinue OAC due to other medical conditions requiring chronic OAC therapy).
3. The subject is deemed by the treating physician to be unsuitable for chronic anticoagulation and/or aspirin therapy due to bleeding risk, allergy, or other reasons.
4. The subject had or is planning to have any cardiac or major non-cardiac interventional or surgical procedure (excluding non-valvular AF ablation and cardioversion) within 30 days prior to or 60 days after randomization [including, but not limited to: percutaneous coronary intervention (PCI), other cardiac ablation (VT ablation, etc.), etc.].
5. The subject had a stroke or transient ischemic attack (TIA) within the 60 days prior to randomization.
6. The subject had a prior major bleeding event per ISTH definition within the 14 days prior to randomization. Lack of resolution of related clinical sequelae, or planned and pending interventions to resolve bleeding/bleeding source, are a further exclusion regardless of timing of the bleeding event.
7. The subject has had a myocardial infarction (MI) documented in the clinical record as either a non-ST elevation MI (NSTEMI) or as an ST-elevation MI (STEMI), with or without intervention, within 90 days prior to randomization.
8. The subject has a history of atrial septal repair or has an ASD/PFO device.
9. The subject has an implanted mechanical valve prosthesis in any position.
10. The subject is of childbearing potential and is, or plans to become pregnant during the time of the study (method of assessment upon study physician's discretion)
11. The subject has a documented life expectancy of less than two years.
12. The subject has a cardiac tumor.
13. The subject has signs/symptoms of acute or chronic pericarditis.
14. There is evidence of tamponade physiology.
15. Contraindications (anatomical or medical) to percutaneous catheterization procedures.
16. The subject has documented NYHA Class IV heart failure.
17. The subject has documented surgical closure of the left atrial appendage.
18. The subject has an active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oussama Wazni, MD, Principal Investigator — The Cleveland Clinic
Locations (114):
- United States (81):
  - Grandview Medical Center, Birmingham, Alabama
  - Heart Center Research, Huntsville, Alabama
  - Alaska Regional Hospital, Anchorage, Alaska
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - Heart Clinic Arkansas, Little Rock, Arkansas
  - Mills Peninsula Health Services, Burlingame, California
  - Scripps Memorial Hospital, La Jolla, California
  - Marin General Hospital, Larkspur, California
  - University of Southern California Hospital, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente Santa Clara Medical Center, Santa Clara, California
  - Marian Regional Medical Center, Santa Maria, California
  - Memorial Hospital, Colorado Springs, Colorado
  - Centura Health, Littleton, Colorado
  - Medical Center of the Rockies (Loveland), Loveland, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - AdventHealth Ocala, Ocala, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - St. Alphonsus Regional Medical Center, Boise, Idaho
  - St. Lukes Idaho Cardiology Associates, Boise, Idaho
  - Edward Hospital, Naperville, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Methodist Hospital of Indianapolis, Indianapolis, Indiana
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - Overland Park Regional Medical Center, Kansas City, Kansas
  - University of Kansas Hospital, Kansas City, Kansas
  - Kansas City Cardiac Arrhythmia Research, Overland Park, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic Hospital, Burlington, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Mercy Research, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Catholic Medical Center, Manchester, New Hampshire
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Northwell Health, Bay Shore, New York
  - New York University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Lindner Center for Research and Education at Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OhioHealth Research and Innovation Institute - Riverside Methodist Hospital, Columbus, Ohio
  - Pinnacle Health at Harrisburg Hospital, Harrisburg, Pennsylvania
  - Presbyterian University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Centennial Medical Center, Nashville, Tennessee
  - Saint Thomas Health, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - HeartPlace Mid-Cities EP, Bedford, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Cardiology Clinic of San Antonio, San Antonio, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - St. Mark's Hospital, Salt Lake City, Utah
  - Chippenham Medical Center, Richmond, Virginia
  - CHI Franciscan Health System, Tacoma, Washington
  - PeaceHealth Southwest Medical, Vancouver, Washington
  - Monongalia General Hospital, Morgantown, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
- Australia (2):
  - Advara HeartCare, Brisbane, Queensland
  - Monash Health, Clayton, Victoria
- Onze Lieve Vrouw Ziekenhuis, Aalst, East Flanders, Belgium
- Aarhus University Hospital, Aarhus, Denmark
- France (8):
  - CHRU de Lille, Lille, Hauts-de-France
  - CHRU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble - Hopital Michallon, Grenoble
  - Hospital Europeen Georges-Pompidou, Paris
  - Clinique Pasteur, Toulouse
  - Centre Hôpital Universitaire Rangueil, Toulouse
  - CHU Henri Mondor, Créteil, Île-de-France Region
  - Hospital de la Pitie-Salpetriere, Paris, Île-de-France Region
- Germany (11):
  - DHZC - Deutsches Herzzentrum der Charité, Berlin
  - Klinik für Kardiologie, Angiologie und Intensivmedizin Mittelallee, Berlin
  - Klinikum Coburg GmbH, Coburg
  - St.Johann Nepomuk Katholisches Hospitalvereinigung Thüringen GmbH, Erfurt
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Universitatsklinik Greifswald, Greifswald
  - Asklepios Klinik Saint Georg, Hamburg
  - Allgemeines Krankenhaus Altona, Hamburg
  - Klinikum St. Georg, Leipzig
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
  - St. Josefs-Hospital GmbH, Wiesbaden
- Italy (2):
  - Centro Cardiologico Monzino, Milan
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino
- St. Antonius Ziekenhuis, Nieuwegein, Utrecht, Netherlands
- Poznan University of Medical Sciences, Poznan, Poland
- Spain (6):
  - Hospital General Universitario, Alicante
  - Hospital Puerta Del Mar, Cadiz
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clinico Salamanca, Salamanca
  - Clinico de Valladolid, Valladolid
  - Hospital Alvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: Yes
URL: http://www.bostonscientific.com/content/gwc/en-US/data-sharing-requests.html

REFERENCES:
- [Derived] Wazni OM, Saliba WI, Nair DG, Marijon E, Schmidt B, Hounshell T, Ebelt H, Skurk C, Oza S, Patel C, Kanagasundram A, Sadhu A, Sundaram S, Osorio J, Mark G, Gupta M, DeLurgio DB, Olson J, Nielsen-Kudsk JE, Boersma LVA, Healey JS, Phillips KP, Asch FM, Wolski K, Roy K, Christen T, Sutton BS, Stein KM, Reddy VY; OPTION Trial Investigators. Left Atrial Appendage Closure after Ablation for Atrial Fibrillation. N Engl J Med. 2025 Apr 3;392(13):1277-1287. doi: 10.1056/NEJMoa2408308. Epub 2024 Nov 16. PMID 39555822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1600 subjects were randomized from 11-Jun-2019 to 16-Jul-2021
Pre-assignment Details: 803 subjects were randomized to the WATCHMAN FLX DEVICE and 797 subjects were randomized to the OAC Control group (ITT analysis set)
Groups:
- Oral Anticoagulant (Control): Catheter ablation for atrial ablation followed by market-approved OAC for the duration of the trial
- WATCHMAN FLX DEVICE: Catheter ablation for atrial fibrillation followed by WATCHMAN FLX Device implant with market-approved OAC and aspirin until the 3-month visit followed by aspirin until at least the 12-month visit
Period: Overall Study
Arm/Group | Oral Anticoagulant (Control) | WATCHMAN FLX DEVICE
Started | 797 | 803
Completed (36-months post-randomization) | 679 | 714
Not Completed | 118 | 89
Not completed — Death | 34 | 29
Not completed — Death > 1095 day (not included in endpoint analyses) | 1 | 2
Not completed — Lost to Follow-up | 28 | 17
Not completed — Physician Decision | 5 | 4
Not completed — Withdrawal by Subject | 43 | 28
Not completed — Reason not reported | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Anticoagulant (Control) | WATCHMAN FLX DEVICE | Total
Number analyzed (Participants) | 797 | 803 | 1600
Age, Continuous [Mean (Standard Deviation); unit: Years at time of Consent] | 69.4 (7.9) | 69.7 (7.4) | 69.5 (7.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 533 | 520 | 1053
  Female | 263 | 283 | 546
  Intersex | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 1 | 2 | 3
  Asian | 1 | 4 | 5
  Black, of African heritage | 11 | 14 | 25
  Caucasian | 686 | 673 | 1359
  Hispanic or Latino | 12 | 13 | 25
  Other | 3 | 3 | 6
  Not disclosed | 83 | 94 | 177
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 562 | 560 | 1122
  Australia | 12 | 10 | 22
  Belgium | 6 | 7 | 13
  Denmark | 13 | 12 | 25
  France | 61 | 66 | 127
  Germany | 100 | 104 | 204
  Italy | 4 | 3 | 7
  Netherlands | 6 | 6 | 12
  Poland | 9 | 8 | 17
  Spain | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint: Stroke, All Cause Death, and Systemic Embolism
Description: Occurrence of stroke (including ischemic and/or hemorrhagic), all cause death, and systemic embolism events adjudicated by an Independent Clinical Event Committee
Time Frame: From randomization to 1095 days post randomization
Population: The primary analysis for the primary effectiveness endpoint was performed on an intent-to-treat basis, with all randomized subjects analyzed as part of their randomized group regardless of the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Anticoagulant (Control) | WATCHMAN FLX DEVICE
Number analyzed (Participants) | 797 | 803
Participants | 44 | 41

2. Primary Outcome: Primary Safety Endpoint: Non-procedural Bleeding
Description: Occurrence of non-procedural bleeding (ISTH major bleeding and clinically relevant non-major bleeding) events adjudicated by an Independent Clinical Event Committee
Time Frame: Non-procedural events are those occurring after 3 days, calculated from implant or attempted implant date for Device patients and from date of randomization for Control patients
Population: The primary analysis for the primary safety endpoint was performed on an intent-to-treat basis, with all randomized subjects analyzed as part of their randomized group regardless of the actual treatment received
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Anticoagulant (Control) | WATCHMAN FLX DEVICE
Number analyzed (Participants) | 797 | 803
Participants | 137 | 65

3. Secondary Outcome: ISTH Major Bleeding
Description: Occurence of ISTH major bleeding (including procedural bleeding) events adjudicated by an Independent Clinical Event Committee
Time Frame: From randomization to 1095 days post randomization
Population: The primary analysis for the secondary endpoint was performed on an intent-to-treat basis, with all randomized subjects analyzed as part of their randomized group regardless of the actual treatment received
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Anticoagulant (Control) | WATCHMAN FLX DEVICE
Number analyzed (Participants) | 797 | 803
Participants | 38 | 30

ADVERSE EVENTS:
Time Frame: Study events reported below include all events that were reported through study completion, up to 3 years. Note: primary endpoint analyses only included deaths that occurred between randomization and 1095 days post-randomization
Description: Site reported
Arm/Group | Oral Anticoagulant (Control) | WATCHMAN FLX DEVICE
All-Cause Mortality (participants affected / at risk) | 35/797 | 31/803
Serious Adverse Events (participants affected / at risk) | 797/797 | 803/803
Other Adverse Events (participants affected / at risk) | 248/797 | 254/803
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Anticoagulant (Control) (N=797) | WATCHMAN FLX DEVICE (N=803)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 3 (3)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 3 (4)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 7 (8) | 9 (9)
Angina pectoris (Cardiac disorders) | 13 (13) | 10 (11)
Angina unstable (Cardiac disorders) | 4 (4) | 5 (5)
Aortic valve disease (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 3 (3) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 125 (176) | 137 (186)
Atrial flutter (Cardiac disorders) | 28 (29) | 35 (47)
Atrial tachycardia (Cardiac disorders) | 9 (9) | 13 (13)
Atrial thrombosis (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 2 (2)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 5 (5) | 6 (6)
Cardiac arrest (Cardiac disorders) | 4 (4) | 3 (3)
Cardiac failure (Cardiac disorders) | 14 (16) | 16 (18)
Cardiac failure acute (Cardiac disorders) | 5 (5) | 9 (9)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 7 (9) | 15 (17)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 16 (18) | 17 (17)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 2 (2)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 2 (2)
Mitral valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 7 (9) | 3 (3)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 4 (4) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 6 (6)
Pericardial haemorrhage (Cardiac disorders) | 1 (2) | 1 (1)
Pericarditis (Cardiac disorders) | 3 (3) | 3 (3)
Sinus arrest (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 7 (7) | 8 (8)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 7 (8) | 4 (5)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 3 (3) | 3 (3)
Tachycardia induced cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 3 (6) | 3 (3)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 7 (7) | 6 (7)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 4 (4)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperaldosteronism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Diplopia (Eye disorders) | 3 (3) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Ocular retrobulbar haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocele (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastritis alcoholic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (14) | 7 (7)
Haematemesis (Gastrointestinal disorders) | 3 (4) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 6 (6)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 8 (9) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Retroperitoneal mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 4 (5)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 2 (2) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 5 (5) | 3 (3)
Cyst (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 3 (3)
Device related thrombosis (General disorders) | 1 (1) | 3 (3)
Drug intolerance (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Medical device site haematoma (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 11 (11) | 6 (8)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumobilia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 3 (3)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 5 (5) | 5 (6)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Corona virus infection (Infections and infestations) | 3 (3) | 6 (6)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 3 (4) | 2 (3)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis listeria (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 20 (25) | 28 (31)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 5 (5)
Septic shock (Infections and infestations) | 4 (4) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 4 (5)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Lumbar puncture (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 (20) | 15 (18)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angioimmunoblastic T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign cardiac neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endocrine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 5 (5)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 5 (5)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 3 (3)
Facial paralysis (Nervous system disorders) | 2 (2) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 7 (8) | 9 (9)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 7 (7) | 11 (11)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 3 (3)
Device failure (Product Issues) | 0 (0) | 1 (1)
Device lead damage (Product Issues) | 1 (1) | 1 (1)
Device leakage (Product Issues) | 0 (0) | 1 (1)
Device loosening (Product Issues) | 0 (0) | 1 (1)
Lead dislodgement (Product Issues) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Mental status changes (Psychiatric disorders) | 3 (3) | 1 (1)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 13 (14) | 15 (19)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 10 (11) | 7 (7)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Urogenital haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penile haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (8)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (6)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 0 (0) | 1 (2)
Medical device change (Surgical and medical procedures) | 1 (1) | 0 (0)
Tricuspid valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Air embolism (Vascular disorders) | 0 (0) | 2 (2)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2) | 2 (3)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 4 (4) | 3 (3)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 5 (7)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 8 (8) | 4 (4)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 4 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (3)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 2 (3) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 4 (4) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 2 (2)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Anticoagulant (Control) (N=797) | WATCHMAN FLX DEVICE (N=803)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 54 (62) | 71 (88)
Atrial flutter (Cardiac disorders) | 21 (24) | 17 (20)
Atrial septal defect acquired (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 6 (6) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac amyloidosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 3 (3)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 4 (4) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3) | 11 (11)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 3 (3)
Conjunctival haemorrhage (Eye disorders) | 6 (6) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 1 (1)
Eyelid haematoma (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Faeces discoloured (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 4 (4) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 5 (5) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site bruise (General disorders) | 1 (1) | 2 (2)
Catheter site haematoma (General disorders) | 1 (1) | 5 (5)
Catheter site haemorrhage (General disorders) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 4 (4)
Chest pain (General disorders) | 6 (6) | 2 (3)
Device related thrombosis (General disorders) | 1 (1) | 11 (12)
Fatigue (General disorders) | 2 (3) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Mass (General disorders) | 0 (0) | 1 (1)
Medical device site haematoma (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 5 (5)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Corona virus infection (Infections and infestations) | 6 (6) | 8 (8)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (5)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 7 (7) | 7 (7)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (2) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Phrenic nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Retinal migraine (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 5 (5)
Transient ischaemic attack (Nervous system disorders) | 5 (5) | 3 (3)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Device electrical impedance issue (Product Issues) | 1 (1) | 0 (0)
Device failure (Product Issues) | 0 (0) | 1 (1)
Device leakage (Product Issues) | 0 (0) | 7 (7)
Lead dislodgement (Product Issues) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4)
Haematuria (Renal and urinary disorders) | 17 (19) | 11 (11)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 2 (2)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 35 (41) | 10 (11)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Vascular purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Atrial appendage closure (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 12 (12) | 5 (5)
Haemorrhage (Vascular disorders) | 5 (5) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Venous haemorrhage (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study had several exclusion criteria and results may not be applicable to the excluded populations. Pulsed field ablation was not available at the time of the trial. Although type of ablation technology used is unlikely to affect antithrombotic strategy, any unique considerations for this ablation method could not be investigated in the present study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT03795298/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT03795298/SAP_001.pdf